CLINICAL TRIAL: NCT03529019
Title: Perioperative Nutritional Optimization in Patients With Critical Limb Ischemia
Brief Title: Nutrition in Patient With Critical Limb Ischemia
Acronym: NutriVasc
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Vascular & Endovascular Surgery Society (Unknown); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H-37324
Record Dates: First submitted 2018-04-13; First posted 2018-05-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Critical Limb Ischemia; Malnutrition; Nutritional Supplements
Keywords: Enhanced Recovery After Surgery Protocol
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Malnutrition

STUDY DESIGN:
Intervention Model Description: Potential subjects with potential malnutrition and critical limb ischemia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nutritional Supplement (Experimental): Administration of Ensure Surgery Immunonutrition Shake and ensure Enlive Advanced Nutrition Shake.
  Interventions: Drug: Ensure Surgery Immunonutrition Shake; Drug: Ensure Enlive Advanced Nutrition Shake

INTERVENTIONS:
Drug: Ensure Surgery Immunonutrition Shake — An FDA approved nutritional supplement. Prepackaged product designed to be administered one week prior to and one week post surgical procedures.
Drug: Ensure Enlive Advanced Nutrition Shake — An FDA approved nutritional supplement. Prepackaged product designed to be administered 2 weeks prior to and 2 weeks post surgical procedure for a period of one week. .

SUMMARY:
A prospective pilot study examining nutritional supplements among vascular surgery patients with Critical Limb Ischemia (CLI). CLI patients have a high rate of malnutrition and has the potential to benefit greatly from nutritional intervention. The investigators plan to evaluate nutrition and functional status of patients by assessing objective lab values and the use of the hand grip strength test. Providing perioperative nutritional supplements to patients has potentially improved their nutritional status, which in turn may improve the patient's clinical status after surgery.

DETAILED DESCRIPTION:
Malnutrition continues to be a considerable public health issue in the United States and is known to be associated with negative health outcomes. Surgeons and hospitals have adopted preoperative nutritional screening and perioperative nutritional supplementation as best practice for modern treatment of general surgery patients. Nutritional optimization has been shown to improve outcomes in these patients and has become integrated as a key component of the Enhanced Recovery After Surgery (ERAS) protocol. Although much progress has been made towards optimizing perioperative nutritional status for general surgery patients in an effort to improve surgical outcomes, there remains a dearth of information on the association between nutritional status and health outcomes after vascular surgery interventions. Recent research has found that up to 50% of general and gastrointestinal surgical patients suffered from malnutrition in the preoperative phase. This finding has led to efforts to optimize the nutritional status of general and gastrointestinal surgery patients in the perioperative phase. Perioperative nutritional supplementation has been shown to reduce morbidity and mortality in various subsets of surgical patients. This research has fallen short of examining nutritional status and outcomes among vascular surgery patients. Published data in this area has been limited to analyses of existing retrospective datasets. Additionally, nutritional research that includes data from vascular surgery patients has been limited to an examination of pre- and post-operative albumin levels in an attempt to find a correlation between these levels and outcomes. Though this research is limited, it has shown that vascular surgery patients with low (<3.5 g/dl) pre-operative albumin levels and critical limb ischemia (CLI) are at increased risk for perioperative morbidity and mortality after lower extremity bypass than vascular surgery patients with high pre-operative albumin levels (>3.5 g/dl). As serum albumin levels can be altered in the acute phase due to inflammation, this research, while valuable, only represents a single component required for the assessment of nutritional status.

Approximately 45.5% patients with CLI have been shown to have signs of preoperative malnutrition when undergoing infrainguinal bypass. Malnutrition remains an underrepresented area of perioperative management for vascular surgery patients. Research on the association between nutritional supplementation and improved vascular surgery outcomes has the potential to enhance the success of lower extremity interventions by validating an optimal adjunctive medical therapy. Patients with CLI in general are at significantly higher risk for perioperative morbidity and resource utilization when compared to other hospitalized patients. Unlike many gastrointestinal surgery patients, these patients often do not have a primary gastrointestinal pathology contributing to their malnutrition; more likely, it may be the result of their comorbidities and an overall failure to thrive. Perioperative nutritional supplementation has the potential to improve the nutritional status of these patients and ultimately improve outcomes. Yet, to date, no prospective trial of nutritional supplementation in CLI patients has been performed.

A multidisciplinary team including nutritionists, vascular surgeons, and surgical critical care surgeons with expertise in perioperative nutrition research has been assembled to conduct a pilot research study examining the impact of nutritional supplementation on vascular surgery outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Critical Limb Ischemia

Exclusion Criteria:

* Female patients who are pregnant or lactating
* Chronic Kidney Disease Stages 4 and 5
* Patients who are on dialysis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in serum albumin levels | baseline and 30 days
  Albumin is a carbohydrate-free protein, which constitutes 55% to 65% of total plasma protein. Albumin results can reflect the nutritional status of the body and other problems with the kidney or liver. A normal albumin range is 3.4 to 5.4 g/dL. Albumin levels will be tested on blood samples on each participant obtained at baseline and 30 days after nutritional supplementation. Lower albumin levels are associated with malnutrition
Change in prealbumin levels | baseline and 30 days
  Prealbumin is a protein produced by the liver and levels can reflect nutritional status. Normal results for a prealbumin blood test for adults are 15 to 36 milligrams per deciliter (mg/dL). Prealbumin levels will be tested on blood samples on each participant obtained at baseline and 30 days after nutritional supplementation. Lower levels of prealbumin are associated with malnutrition.
Change in transferrin levels | baseline and 30 days
  Transferrin is the main protein in the blood that binds to iron and transports it throughout the body. The normal range for transferrin is 170 to 370 mg/dl. Transferrin levels will be tested on blood samples on each participant obtained at baseline and 30 days after nutritional supplementation. Transferrin levels rise with iron deficiency and fall in cases of iron overload.
Change in C-reactive protein levels | baseline and 30 days
  C-reactive protein (CRP) is a substance produced by the liver that increases in the presence of inflammation in the body. C-reactive protein levels will be tested on blood samples on each participant obtained at baseline and 30 days after nutritional supplementation. Lower levels are favorable.

SECONDARY OUTCOMES:
Change in Hand grip strength | baseline and 30 days
  A hand dynamometer will be used to measure hand grip strength. Higher values are favorable.

OTHER OUTCOMES:
Change in ERAS (Enhanced Recovery After Surgery) Malnutrition Screening Test (MST) Scores | baseline and 30 days
  The ERAS Malnutrition Screening Test (MST) is a 3 question survey used to evaluate patient's nutritional status. The 3 questions ask about recent weight loss without trying, amount of the weight loss, and whether eating poorly because of a decreased appetite. Scores of 2 or greater indicate risk of malnutrition. Lower scores are favorable.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Siracuse, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kubota K, Kuroda J, Yoshida M, Okada A, Deguchi T, Kitajima M. Preoperative oral supplementation support in patients with esophageal cancer. J Nutr Health Aging. 2014 Apr;18(4):437-40. doi: 10.1007/s12603-014-0018-2. PMID 24676327
- [Background] Lidder P, Thomas S, Fleming S, Hosie K, Shaw S, Lewis S. A randomized placebo controlled trial of preoperative carbohydrate drinks and early postoperative nutritional supplement drinks in colorectal surgery. Colorectal Dis. 2013 Jun;15(6):737-45. doi: 10.1111/codi.12130. PMID 23406311
- [Background] Kobayashi D, Ishigure K, Mochizuki Y, Nakayama H, Sakai M, Ito S, Kojima H, Kajikawa M, Ando M, Kodera Y. Multi-institutional prospective feasibility study to explore tolerability and efficacy of oral nutritional supplements for patients with gastric cancer undergoing gastrectomy (CCOG1301). Gastric Cancer. 2017 Jul;20(4):718-727. doi: 10.1007/s10120-016-0668-3. Epub 2016 Nov 24. PMID 27885538
- [Background] Short V, Atkinson C, Ness AR, Thomas S, Burden S, Sutton E. Patient experiences of perioperative nutrition within an Enhanced Recovery After Surgery programme for colorectal surgery: a qualitative study. Colorectal Dis. 2016 Feb;18(2):O74-80. doi: 10.1111/codi.13245. PMID 26682875
- [Background] Makuuchi R, Sugisawa N, Kaji S, Hikage M, Tokunaga M, Tanizawa Y, Bando E, Kawamura T, Terashima M. Enhanced recovery after surgery for gastric cancer and an assessment of preoperative carbohydrate loading. Eur J Surg Oncol. 2017 Jan;43(1):210-217. doi: 10.1016/j.ejso.2016.07.140. Epub 2016 Aug 10. PMID 27554250
- [Background] Braga M, Gianotti L, Nespoli L, Radaelli G, Di Carlo V. Nutritional approach in malnourished surgical patients: a prospective randomized study. Arch Surg. 2002 Feb;137(2):174-80. doi: 10.1001/archsurg.137.2.174. PMID 11822956
- [Background] Hughes K, Boyd C, Oyetunji T, Tran D, Chang D, Rose D, Siram S, Cornwell E 3rd, Obisesan T. Racial/ethnic disparities in revascularization for limb salvage: an analysis of the National Surgical Quality Improvement Program database. Vasc Endovascular Surg. 2014 Jul-Aug;48(5-6):402-5. doi: 10.1177/1538574414543276. Epub 2014 Jul 30. PMID 25080452
- [Background] Cerantola Y, Grass F, Cristaudi A, Demartines N, Schafer M, Hubner M. Perioperative nutrition in abdominal surgery: recommendations and reality. Gastroenterol Res Pract. 2011;2011:739347. doi: 10.1155/2011/739347. Epub 2011 May 22. PMID 21687620
- [Background] Leandro-Merhi VA, de Aquino JL, Sales Chagas JF. Nutrition status and risk factors associated with length of hospital stay for surgical patients. JPEN J Parenter Enteral Nutr. 2011 Mar;35(2):241-8. doi: 10.1177/0148607110374477. Epub 2010 Oct 22. PMID 20971940
- [Background] Pirlich M, Schutz T, Norman K, Gastell S, Lubke HJ, Bischoff SC, Bolder U, Frieling T, Guldenzoph H, Hahn K, Jauch KW, Schindler K, Stein J, Volkert D, Weimann A, Werner H, Wolf C, Zurcher G, Bauer P, Lochs H. The German hospital malnutrition study. Clin Nutr. 2006 Aug;25(4):563-72. doi: 10.1016/j.clnu.2006.03.005. Epub 2006 May 15. PMID 16698132